CLINICAL TRIAL: NCT00892177
Title: Phase I/Randomized Phase II Double Blind Study of Either Dasatinib or Placebo Combined With Bevacizumab in Recurrent Glioblastoma
Brief Title: Dasatinib and Bevacizumab in Treating Patients With Recurrent or Progressive High-Grade Glioma or Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-N0872; NCI-2011-01921 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000641746 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Glioblastoma Multiforme
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult mixed glioma; recurrent adult brain tumor; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult anaplastic astrocytoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms; Oligodendroglioma; Astrocytoma | interventions — Bevacizumab; Dasatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive bevacizumab on Day 1 and dasatinib on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: dasatinib
- Arm II (Active Comparator): Patients receive bevacizumab on Day 1 and placebo on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: placebo

INTERVENTIONS:
Biological: bevacizumab — Given intravenously
Drug: dasatinib — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also block the growth of the tumor by blocking blood flow to the tumor. It is not yet known whether bevacizumab together with dasatinib are more effective than a placebo in treating patients with recurrent or progressive high-grade glioma or glioblastoma multiforme.

PURPOSE: This randomized phase I/II trial (Phase I completed) is studying the side effects and best dose of dasatinib when given together with bevacizumab and to see how well it works compared to placebo in treating patients with recurrent or progressive high-grade glioma or glioblastoma multiforme.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter, phase I, dose-escalation study (Phase I completed) of dasatinib followed by a phase II randomized study. Patients are grouped according to study (1 vs 2). Patients in the phase II portion are stratified according to age (> 70 years of age vs ≤ 70 years of age), and ECOG performance status (0 vs 1 or 2).

Phase I: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oral dasatinib once or twice daily on days 1-14 until the maximum-tolerated dose (MTD) is determined. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. (Phase I completed) Please see the Arms section for the Phase II treatment regimens.

OBJECTIVES:

PRIMARY OBJECTIVES:

1. Determine the maximum tolerated dose (MTD) of dasatinib in combination with bevacizumab in high grade glioma patients. (Phase I)
2. To assess the safety and adverse events of the dasatinib in combination with bevacizumab in this patient population. (Phase I)
3. To estimate the efficacy of the bevacizumab combination with dasatinib in recurrent glioblastoma multiforme as measured by progression free survival at six months and compare it with the efficacy of bevacizumab alone. (Phase II)

SECONDARY OBJECTIVES:

1. To describe the overall toxicity associated with the dasatinib/bevacizumab combination. (Phase I)
2. To describe any preliminary evidence of antitumor activity. (Phase I)
3. To assess the time to disease progression. (Phase II)
4. To assess the safety and toxicity of the bevacizumab combination with dasatinib in this patient population. (Phase II)
5. To estimate the efficacy of the bevacizumab combination with dasatinib in recurrent glioblastoma multiforme as measured by overall survival time and compare it with the efficacy of bevacizumab alone. (Phase II)
6. To assess the impact of the treatment on the patient's quality of life (QOL) using the overall score from the FACT-Br (Phase II)

ELIGIBILITY:
Patient Eligibility:

I. Pre-registration:

1. Central pathology review submission. This review is mandatory prior to registration to confirm eligibility.

II. Registration Inclusion Criteria:

1. ≥18 years of age
2. Study 1: Histologic confirmation of grade 3 or 4 glioma, including astrocytoma, oligodendroglioma, and mixed gliomas, as determined by pre-registration central pathology review.
3. Study 2: Histological confirmation of glioblastoma multiforme (grade 4 astrocytoma) as determined by pre-registration central pathology review. NOTE: Variant gliosarcomas are eligible
4. Evidence of tumor progression by MRI or CT scan following RT or following the most recent anti-tumor therapy. Patients who had surgical treatment at recurrence are eligible if there is imaging evidence of disease progression as compared to the first postoperative scan.
5. Bidimensionally measurable or evaluable disease by MRI or CT scan.
6. ECOG Performance Status (PS) 0, 1, or 2.
7. Patient willing to discontinue use of aspirin or medications that inhibit platelet function ≥ 1 week prior to registration.
8. Previous RT and ≥12 weeks since the completion of RT prior to registration.
9. The following laboratory values obtained ≤ 21 days prior to registration.

   * ANC ≥1500
   * PLT ≥100,000
   * Hgb >9.0 g/dL
   * T. bili ≤1.5 x ULN
   * SGOT (AST) ≤ 3 x ULN
   * Creatinine ≤ ULN
10. UPC ratio <1. NOTE: Urine protein must be screened by urine analysis for Urine Protein Creatinine (UPC) ratio. For UPC ratio ≥1.0, 24-hour urine protein must be obtained and the level should be <1000 mg
11. Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
12. Ability to complete questionnaire(s) by themselves or with assistance.
13. Provide informed written consent
14. Willingness to return to enrolling institution for follow-up.
15. Patient willing to provide mandatory tissue samples for research purposes
16. Study 1: Any number of prior chemotherapy regimens for recurrent disease. Study 2: Up to 2 prior chemotherapy regimens with ≤1 regimen for recurrent disease.

III. Exclusion Criteria:

1. Pregnant women, nursing women and men or women of childbearing potential who are unwilling to employ adequate contraception during this study and for up to 6 months after bevacizumab treatment has ended. NOTE: bevacizumab and dasatinib are investigational agents whose genotoxic effects on the developing fetus and newborn are unknown.
2. Prior intratumoral therapy, stereotactic radiosurgery, or interstitial brachytherapy.

   EXCEPTION: Separate lesion on MRI which is not part of the previous treatment field, or convincing evidence of recurrent disease, based on biopsy, MRI spectroscopy, or PET scan.
3. Prior treatment with bevacizumab or VEGF-Trap (Aflibercept).
4. Inadequately controlled hypertension (systolic blood pressure of >150 mmHg or diastolic pressure >100 mmHg on anti-hypertensive medications).

   NOTE: Patients with well-controlled hypertension are eligible.
5. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
6. Immunocompromised patients (other than that related to the use of corticosteroids). NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this study.
7. Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or prior surgical procedures affecting absorption) that impairs ability to swallow pills.
8. Receiving therapeutic anticoagulation with Warfarin. NOTE: Prophylactic anticoagulation (i.e., low dose warfarin) of venous or arterial access devices is allowed, provided that INR <1.5. Therapeutic anti-coagulation with low molecular weight heparin is allowed at time of registration.
9. Evidence of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation).
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
12. Other active malignancy ≤3 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma in-situ of the cervix. Note: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer.
13. History of myocardial infarction or unstable angina ≤6 months prior to registration.
14. New York Heart Association (NYHA) classification II, III or IV congestive heart failure.
15. Core biopsy or other minor surgical procedures ≤7 days prior to registration. Note: Placement of a vascular access device is allowed.
16. Major surgical procedure, open biopsy, or significant traumatic injury ≤28 days prior to registration or anticipation of need for major surgical procedure during the course of the study.
17. Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis ≤6 months prior to registration.
18. History of hypertensive crisis or hypertensive encephalopathy.
19. Known hypersensitivity to any of the components of dasatinib or bevacizumab.
20. Serious, non-healing wound, active ulcer, or untreated bone fracture
21. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤6 months prior to registration.
22. Active or recent history of hemoptysis (≥ ½ teaspoon of bright red blood per episode) ≤30 days prior to registration.
23. History of stroke or transient ischemic attack (TIA) ≤6 months prior to registration.
24. Any evidence of CNS hemorrhage on baseline CT or MRI
25. Any of the following Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes ≤7 days prior to registration (patients must discontinue drug 7 days prior to starting dasatinib)

    * Quinidine, procainamide, disopyramide
    * Amiodarone, sotalol, ibutilide, dofetilide
    * Erythromycin, clarithromycin
    * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
    * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
    * Prochlorperazine
26. Diagnosed congenital long QT syndrome
27. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes)
28. Prolonged QTc interval on pre-entry electrocardiogram (>450 msec)
29. Patients may not have any clinically significant cardiovascular disease including the following:

    * Myocardial infarction or ventricular tachyarrhythmia within 6 months.
    * Prolonged QTc ≥ 480 msec (Fridericia correction)
    * Ejection fraction less than institutional normal
    * Major conduction abnormality (unless a cardiac pacemaker is present)

    Note: Patients with any cardiopulmonary symptoms of unknown cause (e.g., shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (ECG) to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator. Patients with underlying cardiopulmonary dysfunction should be excluded from the study.
30. Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
31. Known pleural or pericardial effusion of any grade
32. Concomitant use of H2 blockers or proton pump inhibitors that cannot be discontinued or switched to locally acting agents (i.e. famotidine or omeprazole.)
33. Use of the following Enzyme Inducing Anti-Convulsive (EIAC) medications is prohibited ≤ 7 days prior to registration: carbamazepine (Tegretol®, Tegretol XR®, Carbatrol®), phenytoin (Dilantin®, Phenytek®), fosphenytoin (Cerebyx®), phenobarbital, pentobarbital and primidone (Mysoline®). Note: Many antiepileptic drugs induce hepatic enzymes. Because dasatinib is metabolized by hepatic enzymes, patients taking antiepileptic medications that induce hepatic enzymes (EIACs) are ineligible for this trial. To be eligible for this trial, patients taking EIACs must be switched to non-EIACs ≥ 7 days prior to registration. The following agents are not known to affect dasatinib metabolism and are acceptable for use: valproic acid (Depakote®, Depacon®), gabapentin (Neurontin®), lamotrigine (Lamictal®), topiramate (Topamax®), tiagabine (Gabitril®), zonisamide (Zonegran®), levetiracetam (Keppra®), clonazepam (Klonopin®) and clobazam (Frisium®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Study Chair — Mayo Clinic
Locations (304):
- United States (304):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Palchak David MD, Pismo Beach, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Women's Health - Wichita, Wichita, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers - Adrian, Adrian, Michigan
  - Toledo Clinic Cancer Centers-Adrian, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Sanford Clinic North-Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Frontier Cancer Center and Blood Institutes-Billings, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Healthcare - Sletten Cancer Institute, Great Falls, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Mount Kisco Medical Group at Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Medical Center, New York, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - McLeod Regional Medical Center, Florence, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Derived] Galanis E, Anderson SK, Twohy EL, Carrero XW, Dixon JG, Tran DD, Jeyapalan SA, Anderson DM, Kaufmann TJ, Feathers RW, Giannini C, Buckner JC, Anastasiadis PZ, Schiff D. A phase 1 and randomized, placebo-controlled phase 2 trial of bevacizumab plus dasatinib in patients with recurrent glioblastoma: Alliance/North Central Cancer Treatment Group N0872. Cancer. 2019 Nov 1;125(21):3790-3800. doi: 10.1002/cncr.32340. Epub 2019 Jul 10. PMID 31290996

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 0: Patients receive 5 mg/kg bevacizumab IV over 90 minutes on Day 1 and 50 mg oral dasatinib twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 1: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and 50 mg oral dasatinib twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 2: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and 70 mg oral dasatinib twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 3: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and 100 mg oral dasatinib twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Arm A (Bevacizumab + Dasatinib): Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral dasatinib 100 mg (2 tablets) twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Arm B (Bevacizumab + Placebo): Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral placebo twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Period: Phase I: Dose Level 0
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I: Dose Level 1
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Started | 0 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I: Dose Level 2
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Started | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I: Dose Level 3
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Started | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Started | 0 | 0 | 0 | 0 | 88 | 40
Completed | 0 | 0 | 0 | 0 | 83 | 38
Not Completed | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Ineligible | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Patients receive (either: 5 or 10 mg/kg) bevacizumab IV over 90 minutes on Day 1 and oral dasatinib (either: 50, 70, or 100 mg) twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo) | Total
Number analyzed (Participants) | 16 | 83 | 38 | 137
Age, Continuous [Median (Full Range); unit: years] | 46.5 [28 to 68] | 58 [29 to 79] | 56.5 [18 to 71] | 57 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 28 | 16 | 47
  Male | 13 | 55 | 22 | 90
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 83 | 38 | 137

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities to Determine Maximum Tolerated Dose (MTD) of Dasatinib in Combination With Bevacizumab (Phase I)
Description: The Maximum Tolerated Dose (MTD) will be based on the assessment of dose-limiting toxicities (DLT) during the first 4 weeks of treatment only (i.e., following the first 2 treatment cycles), and will be defined as the dose at which fewer than one-third of patients experience a DLT to study treatment. The MTD is the dose level at which 0/6 or 1/6 patients experience DLT with the next higher dose having at least 2 out of 3 or 2 out of 6 patients encountering DLT.> Three patients will be treated at each dose level, and can be enrolled simultaneously. If one DLT is encountered, an additional 3 patients will be added to that dose level. If at any point two DLTs are encountered within a given dose level, then the MTD has been exceeded and if only three patients have been treated at the next lower dose three more patients are treated at the next lower dose. The number of patients who developed DLTs are reported here by dose level, with the MTD reported in the statistical analysis section.
Time Frame: 14 days
Population: Adverse event information is available for 4 patients on study 1 dose level 1 (with 1 being a MTD replacement due to disease progression prior to completing cycles 1 and 2).
Measure: Number; unit: participants who developed DLTs
Groups:
- Phase I : Dose Level 0: Patients receive 5 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral dasatinib 50 mg twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I : Dose Level 1: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral dasatinib 50 mg twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I : Dose Level 2: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral dasatinib 70 mg twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Phase I : Dose Level 3 Cohort 1; Phase I: Dose Level 3 Cohort 2: Patients receive 10 mg/kg bevacizumab IV over 90 minutes on Day 1 and oral dasatinib 100 mg twice daily on days 1-14. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I : Dose Level 0 | Phase I : Dose Level 1 | Phase I : Dose Level 2 | Phase I : Dose Level 3 Cohort 1 | Phase I: Dose Level 3 Cohort 2
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3
participants who developed DLTs | 0 | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Phase I : Dose Level 0 vs Phase I : Dose Level 1 vs Phase I : Dose Level 2 vs Phase I : Dose Level 3 Cohort 1 vs Phase I: Dose Level 3 Cohort 2; Test type: Superiority or Other; Maximum Tolerated Dose (mg) = 100

2. Primary Outcome: Progression-free Survival at 6 Months (PFS6) (Phase II)
Description: The primary endpoint is the proportion of patients alive and progression-free 6 months after study treatment initiation (PFS6). All eligible consented patients that received treatment will be considered evaluable. Those who die will be considered to have had disease progression unless documented evidence clearly indicates no progression has occurred. PFS6 is defined as the time from start of study therapy to the date of first observation of disease progression or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The PFS6 will be estimated as the number of evaluable patients progression free and still alive at 6 months divided by the total number of evaluable patients. The confidence interval will be calculated according to the Clopper-Pearson Method.
Time Frame: 6 months
Population: All patients that received treatment and were eligible for assessment were included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 83 | 38
proportion of participants | 0.29 [0.19 to 0.39] | 0.18 [0.08 to 0.34]
Statistical Analysis 1: Comparison: Phase II: Arm A (Bevacizumab + Dasatinib) vs Phase II: Arm B (Bevacizumab + Placebo); Test type: Superiority or Other; p = 0.22, Chi-squared, Corrected; Difference = 0.10, 95% CI 2-sided [-0.052 to 0.262] — Difference in proportion

3. Secondary Outcome: Number of Participants With Adverse Events According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 (Phase II)
Description: Adverse events were collected systematically at the end of each cycle and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0. Events are scored as: 1="Mild symptoms", 2= "Moderate", 3="Severe", 4="Life-threatening", and 5="Death". The number of patients reporting a grade 3 or higher event regardless of attribution are summarized here. A complete list of all adverse events reported during treatment can be found in the Adverse Events Section.
Time Frame: Up to 3 years
Population: All Phase II patients treated and evaluated for adverse events are included in this Phase II endpoint analysis.
Measure: Number; unit: participants
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 83 | 38
participants
  Grade 3 Adverse Event | 42 | 23
  Grade 4 Adverse Event | 8 | 2
  Grade 5 Adverse Event | 5 | 3

4. Secondary Outcome: Overall Survival (Phase II)
Description: Survival time is defined to be the length of time from start of study therapy to death due to any cause. All patients meeting the eligibility criteria that have signed a consent form and begun treatment will be considered evaluable for estimation of the survival distribution. The distribution of overall survival for both arms of the study will be estimated using the Kaplan-Meier method, and be compared using log-rank tests.
Time Frame: Up to 3 years
Population: All eligible Phase II patients are included in this Phase II endpoint analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 83 | 38
months | 7.3 [6.2 to 8.7] | 7.9 [6.6 to 11.3]
Statistical Analysis 1: Comparison: Phase II: Arm A (Bevacizumab + Dasatinib) vs Phase II: Arm B (Bevacizumab + Placebo); Test type: Superiority or Other; p = 0.7, Kaplan Meier; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.61 to 1.4]

5. Secondary Outcome: Time-to-disease Progression (Phase II)
Description: Time-to-disease progression is defined as the time from start of study therapy to documentation of disease progression. Patients who die without documentation of progression will be considered to have had tumor progression at the time of death unless there is documented evidence that no progression occurred before death. Patients who fail to return for evaluation after beginning therapy will be censored for progression on the last day of therapy or date last known to be alive, whichever is later. Patients who are still alive and have not progressed will be censored for progression at the time of the last tumor assessment. Patients who experience major treatment violations will be censored for progression on the date the treatment violation occurred. The time-to-progression distribution will be estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: All eligible Phase II patients are included in this Phase II endpoint analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 83 | 38
months | 3.3 [2.79 to 4.6] | 3.5 [2.83 to 4.6]
Statistical Analysis 1: Comparison: Phase II: Arm A (Bevacizumab + Dasatinib) vs Phase II: Arm B (Bevacizumab + Placebo); Test type: Superiority or Other; p = 0.52, Kaplan Meier; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.76 to 1.7]

6. Secondary Outcome: Patient-reported QOL, as Measure by the Functional Assessment of Cancer Therapy-Brain (FACT-Br) (Phase II)
Description: FACT-Br questionnaires were used to assess QOL at every other cycle of treatment (prior to cycles 3, 5, 7, etc.). FACT-Br includes 50 questions used to assess patients' self-assessment in 4 broad categories: Physical, Social/Family, Emotional, and Function Well-being. Scores range from 0="Not at all", 1="A little bit", 2="Somewhat", 3="Quite a bit", 4="Very Much". Higher scores can be interpreted as having higher quality of life. The scores for all 50 questions were summed to give a total score per patient per cycle. Therefore the possible range is from 0 to 200. Below is the reported mean and standard deviation for patients at baseline and during cycles 2, 4, 6, 8, and 10.
Time Frame: Baseline to cycle 10 (20 weeks).
Population: All Phase II patients that began treatment and submitted at least one FACT-Br questionnaire were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 77 | 34
units on a scale
  Cycle 0 | 139.5 (26.2) | 138.3 (22.4)
  Cycle 2: number analyzed (Participants) | 55 | 23
  Cycle 2 | 131.2 (27.9) | 133.5 (23.5)
  Cycle 4: number analyzed (Participants) | 29 | 16
  Cycle 4 | 137.6 (30.1) | 137.4 (23.1)
  Cycle 6: number analyzed (Participants) | 30 | 13
  Cycle 6 | 140.1 (29.0) | 137.7 (25.7)
  Cycle 8: number analyzed (Participants) | 17 | 9
  Cycle 8 | 142.3 (30.2) | 142.8 (31.1)
  Cycle10: number analyzed (Participants) | 12 | 5
  Cycle10 | 142.1 (34.9) | 149.3 (34.4)
Statistical Analysis 1: Comparison: Phase II: Arm A (Bevacizumab + Dasatinib) vs Phase II: Arm B (Bevacizumab + Placebo); Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -0.223 — The estimate is the net difference between Arm A and Arm B total score using information from all cycles. A negative value means that Arm A has a lower quality of life and a positive value means Arm A has a higher reported quality of life

7. Secondary Outcome: Objective Response (Phase II)
Description: Objective response to treatment will be determined by the results of neurological exam and the MRI and/or CT measurement of the tumor at each evaluation as is used for all NCCTG neuro-oncology trials. The percentage of patients in each response category will be summarized, 95% confidence intervals calculated, and rates between the 2 arms will be compared using a Fisher's Exact test. For bi-dimensionally measurable disease, CR: total disappearance of all tumor and that patients be on no corticosteroids or on only adrenal replacement maintenance; PR: ≥ 50% reduction in product of perpendicular diameters of contrast enhancement or mass with no new lesions, and stable or decreasing steroid dosing; PD: >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions; REGR: unequivocal reduction in extent of contrast-enhancement, or a decrease in mass effect, no new lesions (for evaluable disease); SD: failure to qualify for CR, PR,REGR or PD.
Time Frame: Up to 3 years
Population: All eligible Phase II patients are included in this Phase II endpoint analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Number analyzed (Participants) | 83 | 38
percentage of participants
  CR | 2.4 [0.5 to 7.4] | 2.6 [0 to 11.8]
  PR | 2.4 [0.5 to 7.4] | 5.3 [1.1 to 15.3]
  REGR | 10.8 [6.3 to 17.9] | 18.4 [10.1 to 30.9]
  SD | 57.8 [48.8 to 66.4] | 57.9 [44.6 to 70.1]
  PD | 12.0 [7.2 to 19.3] | 5.3 [1.1 to 15.3]
  Missing/Unknown | 14.5 [9.1 to 22.0] | 10.5 [4.4 to 21.9]
Statistical Analysis 1: Comparison: Phase II: Arm A (Bevacizumab + Dasatinib) vs Phase II: Arm B (Bevacizumab + Placebo); Test type: Superiority; p = 0.6325, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events are assessed 21 days prior to registration, prior to each new cycle, and at time of progression, withdrawal or removal from the study up to 3 years from registration.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for expedited adverse event reporting only, beginning July 1, 2011.
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase I: Dose Level 3 | Phase II: Arm A (Bevacizumab + Dasatinib) | Phase II: Arm B (Bevacizumab + Placebo)
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 2/3 | 1/6 | 32/84 | 18/39
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6 | 83/84 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=3) | Phase I: Dose Level 1 (N=4) | Phase I: Dose Level 2 (N=3) | Phase I: Dose Level 3 (N=6) | Phase II: Arm A (Bevacizumab + Dasatinib) (N=84) | Phase II: Arm B (Bevacizumab + Placebo) (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (21)
Intraoperative complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 0 (N=3) | Phase I: Dose Level 1 (N=4) | Phase I: Dose Level 2 (N=3) | Phase I: Dose Level 3 (N=6) | Phase II: Arm A (Bevacizumab + Dasatinib) (N=84) | Phase II: Arm B (Bevacizumab + Placebo) (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (28) | 2 (24) | 2 (22) | 5 (20) | 67 (432) | 14 (38)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 10 (17) | 7 (14)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (6) | 1 (6) | 1 (2) | 3 (13) | 50 (186) | 12 (51)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (6) | 1 (2) | 0 (0) | 11 (17) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (13) | 4 (9)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 31 (82) | 11 (37)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (35) | 4 (6)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (50) | 4 (37) | 3 (29) | 6 (57) | 73 (478) | 35 (241)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 16 (18) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (11) | 1 (1)
Blood gonadotrophin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (14) | 0 (0) | 0 (0) | 0 (0) | 29 (97) | 6 (13)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 13 (35) | 7 (19)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (23) | 0 (0) | 0 (0) | 0 (0) | 14 (51) | 1 (3)
Platelet count decreased (Investigations) | 2 (16) | 1 (1) | 2 (4) | 3 (5) | 47 (180) | 13 (29)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 27 (182) | 11 (105)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (30) | 0 (0) | 0 (0) | 34 (114) | 13 (70)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (14) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 21 (33) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (48) | 2 (7)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (4)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (19)
Acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (12) | 4 (4)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 2 (2)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (22)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 4 (7)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (14) | 3 (14)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (15) | 1 (5)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (14) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (16) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (11) | 2 (4) | 4 (14) | 28 (131) | 18 (92)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes